CLINICAL TRIAL: NCT06903884
Title: A Randomized Controlled Trial of 3% Diquafosol Ophthalmic Solution for Active Moderate-to-Severe Vernal Keratoconjunctivitis
Brief Title: 3% Diquafosol Ophthalmic Solution for Active Moderate-to-Severe Vernal Keratoconjunctivitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VKC001
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: Vernal Keratoconjunctivitis; Dry eye disease; Diquafosol; 0.1% Cyclosporin A
MeSH Terms: conditions — Conjunctivitis, Allergic; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: One group of subjects will receive topical treatment with 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion; another group of subjects will receive 0.1% Cyclosporin A cationic ophthalmic emulsion
Who Masked: Participant, Investigator
Masking Description: It is a double-masked randomized study. Assigned treatment of a specific patients would be kept confidential in both the recruited participants and investigators. To keep the investigators and subjects blind to the study treatment, all investigational drugs are removed from their commercial packaging, wrapped in aluminium foil, double-wrapped in plastic bags, and distributed to participants by an independent clinical research coordinator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion (Experimental): 3% Diquafosol eyedrops 6x/day + 0.1% Cyclosporin A twice a day
  Interventions: Drug: 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion
- 0.1% Cyclosporin A cationic ophthalmic emulsion (Active Comparator): 0.1% Cyclosporin A eyedrops twice a day + preservative free sodium hyaluronate eyedrops 6x/day
  Interventions: Drug: 0.1% Cyclosporin A cationic ophthalmic emulsion

INTERVENTIONS:
Drug: 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion — This arm is to investigate whether patients with moderate-to-severe VKC and keratitis will benefit from the addition of Diquafosol ophthalmic solution
  Arms: 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion
Drug: 0.1% Cyclosporin A cationic ophthalmic emulsion — This arm is a control group to investigate whether patients with moderate-to-severe VKC and keratitis will benefit from the addition of Diquafosol ophthalmic solution
  Arms: 0.1% Cyclosporin A cationic ophthalmic emulsion

SUMMARY:
The aim of the study is to investigate whether patients with moderate-to-severe VKC and keratitis will benefit from the addition of Diquafosol ophthalmic solution in terms of symptoms and signs of VKC, tear film metrics, ocular surface inflammation and quality of life. Potential beneficial effect of Diquafosol treatment on top of current standard use of topical immunosuppressant therapy in VKC would be studied.

Subject at least aged 6 and above with clinical diagnosis of vernal keratoconjunctivitis would be invited to join this study and perform the following assessments:

1. best corrected visual acuity,
2. slit lamp biomicroscope examination,
3. tear meniscus height and non-invasive keratographic tear breakup time(NIKBUT) measurement,
4. cornea fluorescein staining (CFS) and
5. Schirmer's I test. Doctor will prescribe eyedrop, 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion or 0.1% Cyclosporin A cationic ophthalmic emulsion at the end of examination. Subjects will be followed up at 4 weeks, 8 weeks, 16 weeks after treatment.

All participants will be required to answer a standardised questionnaire relating to severity of VKC and dry eye disease.

DETAILED DESCRIPTION:
Aim To compare the four-month clinical efficacy of topical treatment with 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion versus 0.1% Cyclosporin A cationic ophthalmic emulsion in reducing symptoms and signs of active moderate-to-severe vernal keratoconjunctivitis (grade of 2 to 4 on the Bonini severity scale) with keratitis (corneal fluorescein staining score of 1-5 on the modified Oxford scale).

Study design A single-centre prospective double-blinded randomized controlled trial

Hypothesis The addition of topical treatment with 3% Diquafosol ophthalmic solution is superior to 0.1% Cyclosporin cationic ophthalmic emulsion alone in improving symptoms and signs of moderate-to-severe VKC with keratitis at four months of use.

Methods This is a single-centre, prospective, 16-week, randomized, double-blinded controlled clinical trial investigating the clinical efficacy and safety of combined topical treatment with 3% Diquafosol ophthalmic solution and 0.1% Cyclosporin A cationic ophthalmic emulsion and versus topical treatment with 0.1% Cyclosporin A cationic ophthalmic emulsion in patients with moderate-to-severe vernal keratoconjunctivitis and keratitis. The study will also investigate the longitudinal changes in tear cytokines and correlate them with changes in VKC signs and tear film metrics. The study will be performed in accordance with the principles of the Declaration of Helsinki, the International Conference on Harmonization, Good Clinical Practice guidelines, and all applicable laws and regulations. Written informed consent will be obtained from each patient before enrolment in the study. A clinical trials certificate will be obtained from the Department of Health, Hong Kong SAR.

Sample size The study will recruit 94 subjects with moderate-to-severe VKC at eye clinics in Hong Kong West cluster (QMH and GH).

Sample size Calculation Sample size calculation is based on the findings from a prospective study comparing the combined use of 3% Diquafosol and 0.1% Cyclosporin versus 0.1% Cyclosporin alone in the treatment of dry eye disease in 279 subjects [36]. It is anticipated that a similar, if not larger, effective size in VKC patients compared to dry eye patients would be seen. In this study the mean change in cornea staining score between baseline and week 12 was significantly higher in Cyclosporin A and Diquafosol combination therapy (2.91 ± 3.93) than in Cyclosporin A monotherapy (0.93± 2.22). The estimated Cohen's d for this study is approximately 0.620. Based on calculations, approximately 41 participants per group to achieve a study power of 80% with a significance level of 0.05 and the estimated effect size of 0.620 is needed. Considering a 10% dropout rate, the adjusted sample size per group would be approximately 47 participants.

Randomization method Randomisation is conducted by computer-generated random number allocation and will be applied to sequentially enrolled participants. The randomisation schedule is pre-determined, prior to commencing participant recruitment, such that the investigator involved in baseline participant assessment will have no involvement in treatment allocation. Block randomization is performed to ensure 1:1 distribution into treatment groups.

Double-blinding To keep the investigators and subjects blind to the study treatment, all investigational drugs are removed from their commercial packaging, wrapped in aluminium foil, double-wrapped in plastic bags, and distributed to participants by an independent clinical research coordinator.

Rescue Therapy During the study period rescue medication (Loteprednolol 0.5% one drop 4x/day for up to 5 days) is permitted in the event of worsening of ocular surface symptoms. A maximum of 2 courses were allowed between study visits. Any use of rescue therapy is documented in the eyedrop diary and serves as one of the outcome measures.

Patient Workflow The patient workflow is aimed at obtaining clear and comprehensive documentation of symptoms and signs baseline and each subsequent visit after initiation of intervention. Furthermore, documentation of adverse events is achieved via assessment of best corrected visual acuity, intraocular pressure measurement, general periorbital area assessment and slit lamp biomicroscope assessment. See Figure 1. Study Workflow

In particular, the sequence of clinical assessments must be done in order of sequence from least invasive to most invasive, as any touching of the ocular surface or manipulation of the eyelids will stimulate tear secretion. Least invasive tests include imaging-based assessments without manipulation or touching of the ocular surface, include best corrected visual acuity, slit lamp biomicroscope assessment, NIKBUT and tear meniscus height. Mildly invasive tests include those that require gentle touching of the ocular surface, such as fluorescein cornea staining. Moderately invasive tests include those with prolonged ocular surface contact, such as the Schirmer's I test for tear collection

ELIGIBILITY:
Inclusion Criteria:

* Subject at least aged 6 and above
* Clinical diagnosis of vernal keratoconjunctivitis
* Evidence of active moderate-to-severe disease: At least Grade 2 on the Bonini scale of VKC clinical presentation (moderate-to-severe) [38].
* Evidence of keratitis: At least Grade 1 on the Modified Oxford scale for cornea fluorescein staining as reported by Bron et al [39].
* Experienced 1 or more recurrences of VKC during the previous year

Exclusion Criteria:

* Nasolacrimal duct obstruction
* Impaired blinking function
* Active ocular infection or history of ocular herpes, varicella zoster or vaccinia virus infection
* Any ocular disease that would require topical ocular treatment during the study
* Use of cyclosporin A or tacrolimus eyedrops, or use of systemic immunosuppressants within 3 months before enrolment
* Any ocular surgery within 6 months before enrolment

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cornea Fluorescein Staining (CFS) score from baseline to 4 weeks, 8 weeks and 16 weeks between study groups | From baseline to 4 months post- treatment between study groups
  Higher values mean inferior outcomes. Graded according to the modified Oxford grading scale (range 0, 0.5, 1, 2, 3, 4, 5). A difference in score of at least 2 levels (i.e. 4 to 2) or complete resolution of staining (i.e. 0) are both considered clinically significant endpoints.

SECONDARY OUTCOMES:
Percentage of patients requiring rescue topical steroid therapy at 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  Number of patients requiring rescue topical steroid therapy divided by all patients participated in this study
Percentage of patients with improvement in Cornea Fluorescein Staining (CSF) at 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  Number of patients with improvement in CFS requiring rescue topical steroid therapy divided by all patients participated in this study
Change in best corrected visual acuity from baseline to 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  From logmar(1.0 to -0.1)
Change in Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) score from baseline to 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  Range from 0-28, one mark was collected per patient, with higher scores meaning worse
Change in Quality of Life in Children with Vernal Keratoconjunctivitis (QUICK) score from baseline to 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  Range from 0-48, one mark was collected per patient, with higher scores meaning worse outcomes
Change in NIKBUT from baseline to 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  NIKBUT is measured in seconds and average of 3 consecutive readings is taken. Higher values mean better outcomes.
Change in tear meniscus height from baseline to 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  In millimetres. Readings serve as objective parameters for tear volume
Change in tear cytokines from baseline to 4 weeks, 8 weeks and 16 weeks | From baseline to 4 months post- treatment between study groups
  Percentage change in tear cytokines analysis done in lab

OTHER OUTCOMES:
Incidence of ocular adverse events | From baseline to 4 months post- treatment between study groups
  Number of patients with ocular adverse events divided by all patients participated in this study
Incidence of non-ocular adverse events | From baseline to 4 months post- treatment between study groups
  Number of patients with non-ocular adverse events divided by all patients participated in this study
• Incremental cost-effectiveness ratio (ICER) in cost per quality-adjusted life year (QALYs) gained. | From baseline to 4 months post- treatment between study groups
  It is defined by the difference in cost between two possible interventions, divided by the difference in their effect.

CONTACTS AND LOCATIONS:
Overall Officials: Kendrick Co Shih, Principal Investigator — The University of Hong Kong, Grantham Hospital

REFERENCES:
- [Background] Biermann J, Bosche F, Eter N, Beisse F. Treating Severe Pediatric Keratoconjunctivitis with Topical Cyclosporine A. Klin Monbl Augenheilkd. 2022 Nov;239(11):1374-1380. doi: 10.1055/a-1556-1182. Epub 2021 Nov 3. English, German. PMID 34731901
- [Background] Bleik JH, Tabbara KF. Topical cyclosporine in vernal keratoconjunctivitis. Ophthalmology. 1991 Nov;98(11):1679-84. doi: 10.1016/s0161-6420(91)32069-4. PMID 1800929
- [Background] Bremond-Gignac D, Doan S, Amrane M, Ismail D, Montero J, Nemeth J, Aragona P, Leonardi A; VEKTIS Study Group. Twelve-Month Results of Cyclosporine A Cationic Emulsion in a Randomized Study in Patients With Pediatric Vernal Keratoconjunctivitis. Am J Ophthalmol. 2020 Apr;212:116-126. doi: 10.1016/j.ajo.2019.11.020. Epub 2019 Nov 23. PMID 31770513
- [Background] Coban-Karatas M, Ozkale Y, Altan-Yaycioglu R, Sizmaz S, Pelit A, Metindogan S, Canturk-Ugurbas S, Aydin-Akova Y. Efficacy of topical 0.05% cyclosporine treatment in children with severe vernal keratoconjunctivitis. Turk J Pediatr. 2014 Jul-Aug;56(4):410-7. PMID 25818961
- [Background] De Smedt S, Nkurikiye J, Fonteyne Y, Tuft S, De Bacquer D, Gilbert C, Kestelyn P. Topical ciclosporin in the treatment of vernal keratoconjunctivitis in Rwanda, Central Africa: a prospective, randomised, double-masked, controlled clinical trial. Br J Ophthalmol. 2012 Mar;96(3):323-8. doi: 10.1136/bjophthalmol-2011-300415. Epub 2011 Oct 14. PMID 22001151
- [Background] Gupta V, Sahu PK. Topical cyclosporin A in the management of vernal keratoconjunctivitis. Eye (Lond). 2001 Feb;15(Pt 1):39-41. doi: 10.1038/eye.2001.10. PMID 11318292
- [Background] Keklikci U, Dursun B, Cingu AK. Topical cyclosporine a 0.05% eyedrops in the treatment of vernal keratoconjunctivitis - randomized placebo-controlled trial. Adv Clin Exp Med. 2014 May-Jun;23(3):455-61. doi: 10.17219/acem/37145. PMID 24979519
- [Background] Labcharoenwongs P, Jirapongsananuruk O, Visitsunthorn N, Kosrirukvongs P, Saengin P, Vichyanond P. A double-masked comparison of 0.1% tacrolimus ointment and 2% cyclosporine eye drops in the treatment of vernal keratoconjunctivitis in children. Asian Pac J Allergy Immunol. 2012 Sep;30(3):177-84. PMID 23156846
- [Background] Al-Amri AM, Mirza AG, Al-Hakami AM. Tacrolimus Ointment for Treatment of Vernal Keratoconjunctivitis. Middle East Afr J Ophthalmol. 2016 Jan-Mar;23(1):135-8. doi: 10.4103/0974-9233.164616. PMID 26957853
- [Background] Al-Amri AM, Fiorentini SF, Albarry MA, Bamahfouz AY. Long-term use of 0.003% tacrolimus suspension for treatment of vernal keratoconjunctivitis. Oman J Ophthalmol. 2017 Sep-Dec;10(3):145-149. doi: 10.4103/ojo.OJO_232_2014. PMID 29118487
- [Background] Caputo R, Marziali E, de Libero C, Di Grande L, Danti G, Virgili G, Villani E, Mori F, Bacci GM, Lucenteforte E, Pucci N. Long-Term Safety and Efficacy of Tacrolimus 0.1% in Severe Pediatric Vernal Keratoconjunctivitis. Cornea. 2021 Nov 1;40(11):1395-1401. doi: 10.1097/ICO.0000000000002751. PMID 34029239
- [Background] Chatterjee S, Agrawal D. Tacrolimus in Corticosteroid-Refractory Vernal Keratoconjunctivitis. Cornea. 2016 Nov;35(11):1444-1448. doi: 10.1097/ICO.0000000000000918. PMID 27310883
- [Background] Chen M, Wei A, Ke B, Zou J, Gong L, Wang Y, Zhang C, Xu J, Yin J, Hong J. Combination of 0.05% Azelastine and 0.1% Tacrolimus Eye Drops in Children With Vernal Keratoconjunctivitis: A Prospective Study. Front Med (Lausanne). 2021 Sep 17;8:650083. doi: 10.3389/fmed.2021.650083. eCollection 2021. PMID 34604246
- [Background] Fukushima A, Ohashi Y, Ebihara N, Uchio E, Okamoto S, Kumagai N, Shoji J, Takamura E, Nakagawa Y, Namba K, Fujishima H, Miyazaki D. Therapeutic effects of 0.1% tacrolimus eye drops for refractory allergic ocular diseases with proliferative lesion or corneal involvement. Br J Ophthalmol. 2014 Aug;98(8):1023-7. doi: 10.1136/bjophthalmol-2013-304453. Epub 2014 Apr 2. PMID 24695688
- [Background] Heikal MA, Soliman TT, Abousaif WS, Shebl AA. A comparative study between ciclosporine A eye drop (2%) and tacrolimus eye ointment (0.03%) in management of children with refractory vernal keratoconjunctivitis. Graefes Arch Clin Exp Ophthalmol. 2022 Jan;260(1):353-361. doi: 10.1007/s00417-021-05356-0. Epub 2021 Aug 28. PMID 34453603
- [Background] Hirota A, Shoji J, Inada N, Shiraki Y, Yamagami S. Evaluation of Clinical Efficacy and Safety of Prolonged Treatment of Vernal and Atopic Keratoconjunctivitis Using Topical Tacrolimus. Cornea. 2022 Jan 1;41(1):23-30. doi: 10.1097/ICO.0000000000002692. PMID 34870621
- [Background] Kheirkhah A, Zavareh MK, Farzbod F, Mahbod M, Behrouz MJ. Topical 0.005% tacrolimus eye drop for refractory vernal keratoconjunctivitis. Eye (Lond). 2011 Jul;25(7):872-80. doi: 10.1038/eye.2011.75. Epub 2011 Apr 8. PMID 21475312
- [Background] Kumari R, Saha BC, Sinha BP, Mohan N. Tacrolimus versus Cyclosporine- Comparative Evaluation as First line drug in Vernal keratoconjuctivitis. Nepal J Ophthalmol. 2017 Jul;9(18):128-135. doi: 10.3126/nepjoph.v9i2.19257. PMID 29634701
- [Background] Muller GG, Jose NK, de Castro RS. Topical tacrolimus 0.03% as sole therapy in vernal keratoconjunctivitis: a randomized double-masked study. Eye Contact Lens. 2014 Mar;40(2):79-83. doi: 10.1097/ICL.0000000000000001. PMID 24418865
- [Background] Pucci N, Caputo R, di Grande L, de Libero C, Mori F, Barni S, di Simone L, Calvani A, Rusconi F, Novembre E. Tacrolimus vs. cyclosporine eyedrops in severe cyclosporine-resistant vernal keratoconjunctivitis: A randomized, comparative, double-blind, crossover study. Pediatr Allergy Immunol. 2015 May;26(3):256-261. doi: 10.1111/pai.12360. PMID 25712437
- [Background] Samyukta SK, Pawar N, Ravindran M, Allapitchai F, Rengappa R. Monotherapy of topical tacrolimus 0.03% in the treatment of vernal keratoconjunctivitis in the pediatric population. J AAPOS. 2019 Feb;23(1):36.e1-36.e5. doi: 10.1016/j.jaapos.2018.09.010. Epub 2019 Jan 19. PMID 30664932
- [Background] Shoughy SS, Jaroudi MO, Tabbara KF. Efficacy and safety of low-dose topical tacrolimus in vernal keratoconjunctivitis. Clin Ophthalmol. 2016 Apr 7;10:643-7. doi: 10.2147/OPTH.S99157. eCollection 2016. PMID 27103784
- [Background] Wan Q, Tang J, Han Y, Wang D, Ye H. Therapeutic Effect of 0.1% Tacrolimus Eye Drops in the Tarsal Form of Vernal Keratoconjunctivitis. Ophthalmic Res. 2018;59(3):126-134. doi: 10.1159/000478704. Epub 2017 Aug 12. PMID 28803239
- [Background] Zanjani H, Aminifard MN, Ghafourian A, Pourazizi M, Maleki A, Arish M, Shahrakipoor M, Rohani MR, Abrishami M, Khafri Zare E, Barzegar Jalali F. Comparative Evaluation of Tacrolimus Versus Interferon Alpha-2b Eye Drops in the Treatment of Vernal Keratoconjunctivitis: A Randomized, Double-Masked Study. Cornea. 2017 Jun;36(6):675-678. doi: 10.1097/ICO.0000000000001200. PMID 28399035
- [Background] Villani E, Dello Strologo M, Pichi F, Luccarelli SV, De Cilla S, Serafino M, Nucci P. Dry Eye in Vernal Keratoconjunctivitis: A Cross-Sectional Comparative Study. Medicine (Baltimore). 2015 Oct;94(42):e1648. doi: 10.1097/MD.0000000000001648. PMID 26496269
- [Background] Sacchetti M, Baiardini I, Lambiase A, Aronni S, Fassio O, Gramiccioni C, Bonini S, Bonini S. Development and testing of the quality of life in children with vernal keratoconjunctivitis questionnaire. Am J Ophthalmol. 2007 Oct;144(4):557-63. doi: 10.1016/j.ajo.2007.06.028. Epub 2007 Aug 13. PMID 17693381
- [Background] Zhang SY, Li J, Liu R, Lao HY, Fan Z, Jin L, Liang L, Liu Y. Association of Allergic Conjunctivitis With Health-Related Quality of Life in Children and Their Parents. JAMA Ophthalmol. 2021 Aug 1;139(8):830-837. doi: 10.1001/jamaophthalmol.2021.1708. PMID 34110380
- [Background] Leonardi A, Abatangelo G, Cortivo R, Secchi AG. Collagen types I and III in giant papillae of vernal keratoconjunctivitis. Br J Ophthalmol. 1995 May;79(5):482-5. doi: 10.1136/bjo.79.5.482. PMID 7612563
- [Background] Ali A, Bielory L, Dotchin S, Hamel P, Strube YNJ, Koo EB. Management of vernal keratoconjunctivitis: Navigating a changing treatment landscape. Surv Ophthalmol. 2024 Mar-Apr;69(2):265-278. doi: 10.1016/j.survophthal.2023.10.008. Epub 2023 Oct 26. PMID 37890678
- [Background] Nichols KK, Yerxa B, Kellerman DJ. Diquafosol tetrasodium: a novel dry eye therapy. Expert Opin Investig Drugs. 2004 Jan;13(1):47-54. doi: 10.1517/13543784.13.1.47. PMID 14680452
- [Background] Park JH, Moon SH, Kang DH, Um HJ, Kang SS, Kim JY, Tchah H. Diquafosol Sodium Inhibits Apoptosis and Inflammation of Corneal Epithelial Cells Via Activation of Erk1/2 and RSK: In Vitro and In Vivo Dry Eye Model. Invest Ophthalmol Vis Sci. 2018 Oct 1;59(12):5108-5115. doi: 10.1167/iovs.17-22925. PMID 30372737
- [Background] Koh S. Clinical utility of 3% diquafosol ophthalmic solution in the treatment of dry eyes. Clin Ophthalmol. 2015 May 15;9:865-72. doi: 10.2147/OPTH.S69486. eCollection 2015. PMID 26028958
- [Background] Wu D, Chen WQ, Li R, Wang Y. Efficacy and safety of topical diquafosol ophthalmic solution for treatment of dry eye: a systematic review of randomized clinical trials. Cornea. 2015 Jun;34(6):644-50. doi: 10.1097/ICO.0000000000000429. PMID 25909234
- [Background] Sun X, Liu L, Liu C. Topical diquafosol versus hyaluronic acid for the treatment of dry eye disease: a meta-analysis of randomized controlled trials. Graefes Arch Clin Exp Ophthalmol. 2023 Dec;261(12):3355-3367. doi: 10.1007/s00417-023-06083-4. Epub 2023 May 10. PMID 37162564
- [Background] Jeon HS, Hyon JY. The Efficacy of Diquafosol Ophthalmic Solution in Non-Sjogren and Sjogren Syndrome Dry Eye Patients Unresponsive to Artificial Tear. J Ocul Pharmacol Ther. 2016 Sep;32(7):463-8. doi: 10.1089/jop.2015.0081. Epub 2016 Jun 13. PMID 27294831
- [Background] Eom Y, Song JS, Kim HM. Effectiveness of Topical Cyclosporin A 0.1%, Diquafosol Tetrasodium 3%, and Their Combination, in Dry Eye Disease. J Ocul Pharmacol Ther. 2022 Dec;38(10):682-694. doi: 10.1089/jop.2022.0031. PMID 36473191
- [Background] So HR, Baek J, Lee JY, Kim HS, Kim MS, Kim EC. Comparison of matrix metallopeptidase-9 expression following cyclosporine and diquafosol treatment in dry eye. Ann Med. 2023 Dec;55(1):2228192. doi: 10.1080/07853890.2023.2228192. PMID 37354028
- [Background] Bonini S, Bonini S, Lambiase A, Marchi S, Pasqualetti P, Zuccaro O, Rama P, Magrini L, Juhas T, Bucci MG. Vernal keratoconjunctivitis revisited: a case series of 195 patients with long-term followup. Ophthalmology. 2000 Jun;107(6):1157-63. doi: 10.1016/s0161-6420(00)00092-0. PMID 10857837
- [Background] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260